CLINICAL TRIAL: NCT02537119
Title: Massage Therapy on Hamstrings in Patients With Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Fco. Javier Montanez Aguilera, Doctor, Cardenal Herrera University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Cardenal Herrera University
Record Dates: First submitted 2015-06-26; First posted 2015-09-01 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dynamic massage therapy (Experimental): Rubbing on hamstrings combined with articular movement
  Interventions: Procedure: Dynamic massage therapy
- Massage therapy (Active Comparator): Rubbing on hamstrings
  Interventions: Procedure: Massage therapy

INTERVENTIONS:
Procedure: Dynamic massage therapy — Dynamic massage therapy on hamstring combined with knee extension
  Arms: Dynamic massage therapy
Procedure: Massage therapy — Rubbing on hamstrings
  Arms: Massage therapy

SUMMARY:
Effectiveness of a technique of dynamic massage therapy in the hamstrings in patients with nonspecific low back pain.

DETAILED DESCRIPTION:
The main objective of this study is to test the effectiveness of a technique of dynamic massage therapy in the hamstrings in patients with nonspecific low back pain. Secondary objectives are assess whether the technique of dynamic massage therapy increases the extensibility of the hamstrings, assess whether the treatment of hamstrings decreases low back pain and determine whether the application of this technique decreases the disability associated with nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old.
* Low back pain with over three months of evolution.
* Practice sports regularly (at least three times a week).

Exclusion Criteria:

* Fractures, Tumors, congenital anomalies, rheumatic diseases, infectious or inflammatory processes.
* Pathology Nerve root
* Presence of neurological deficit or neuromuscular diseases.
* Surgery
* Physiotherapy treatment for low back pain in the last 30 days.
* Drugs in previous 24h

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Hamstrings extensibility measured with sit-and-reach test | Two weeks
  Fixing a meter stick on top of a solid box so that 26 cm of the ruler extend over the front edge of the box toward the test subject. Used to check the increase in hip flexion.

SECONDARY OUTCOMES:
Low back pain measured with visual analog scale | Two weeks. Participants will be followed for four weeks after completion of the intervention
  The subject indicates the intensity of pain by marking a 100-mm horizontal line with two extremes: no pain and worst imaginable pain. Used to check the decrease low back pain
Low back disability measured with the Oswestry Disability Questionnaire | Two weeks. Participants will be followed for four weeks after completion of the intervention
  Oswestry Disability Questionnaire is an important tool to measure functional low back disability. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated as follows:
  Example: 16 (total scored) 50 (total possible score) x 100 = 32%

CONTACTS AND LOCATIONS:
Overall Officials: FJavier Montañez-Aguilera, Doctor, Principal Investigator — Cardenal Herrera University
Locations (1):
- CEU Cardenal Herrera University, Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pecos-Martin D, Montanez-Aguilera FJ, Gallego-Izquierdo T, Urraca-Gesto A, Gomez-Conesa A, Romero-Franco N, Plaza-Manzano G. Effectiveness of dry needling on the lower trapezius in patients with mechanical neck pain: a randomized controlled trial. Arch Phys Med Rehabil. 2015 May;96(5):775-81. doi: 10.1016/j.apmr.2014.12.016. Epub 2015 Jan 9. PMID 25582412
- [Background] Montanez-Aguilera FJ, Valtuena-Gimeno N, Pecos-Martin D, Arnau-Masanet R, Barrios-Pitarque C, Bosch-Morell F. Changes in a patient with neck pain after application of ischemic compression as a trigger point therapy. J Back Musculoskelet Rehabil. 2010;23(2):101-4. doi: 10.3233/BMR-2010-0255. PMID 20555123
- [Background] Aguilera FJ, Martin DP, Masanet RA, Botella AC, Soler LB, Morell FB. Immediate effect of ultrasound and ischemic compression techniques for the treatment of trapezius latent myofascial trigger points in healthy subjects: a randomized controlled study. J Manipulative Physiol Ther. 2009 Sep;32(7):515-20. doi: 10.1016/j.jmpt.2009.08.001. PMID 19748402